CLINICAL TRIAL: NCT00767403
Title: An Internet Intervention for Childhood Constipation and Encopresis
Brief Title: Internet Intervention for Childhood Encopresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 13846; 5R01HD028160-16 (NIH)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Encopresis
MeSH Terms: conditions — Encopresis

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Internet Intervention + Stepped Care
- 2 (Active Comparator)
  Interventions: Behavioral: Internet Intervention
- 3 (Active Comparator)
  Interventions: Behavioral: Patient Education Website

INTERVENTIONS:
Behavioral: Internet Intervention + Stepped Care — Participants will spend about 1 hour each week for 6 weeks using the Internet Intervention. In the first week, users will complete tutorials covering the three main components of treatment: 1) anatomy, physiology and pathophysiology of digestion; 2) education on clean-out and laxative treatments; and 3) behavioral treatment for encopresis. In subsequent weeks, users will complete weekly "follow-ups," where they answer a series of questions about their progress and needs. The program then assigns additional intervention modules based on the difficulties the participants endorses. The 22 modules target a variety of issues including fears of toilet use; social isolation; administering, adjusting, and tapering laxatives; diet; hygiene; and preventing relapses. In addition to automatic emails, participants in this group will also receive additional support based on whether they complete specific intervention milestones.
  Arms: 1
Behavioral: Internet Intervention — As described in Arm 1 above, participants will spend about 1 hour each week for 6 weeks using the Internet intervention. In the first week, users will complete tutorials covering the three main components of treatment: 1) anatomy, physiology and pathophysiology of digestion; 2) education on clean-out and laxative treatments; and 3) behavioral treatment for encopresis. In subsequent weeks, users will complete weekly "follow-ups," where they answer a series of questions about their progress and needs. The program will then assign additional intervention modules based on the difficulties the participant endorses. The 22 modules target a variety of issues including fears of toilet use; social isolation; administering, adjusting, and tapering laxatives; diet; hygiene; and preventing relapses.
  Arms: 2
Behavioral: Patient Education Website — Participants will be given access to a relevant patient education website. It will contain material on managing and treating the behaviors and symptoms of childhood encopresis.
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness of an Internet intervention designed to reduce the behaviors and symptoms of pediatric encopresis.

DETAILED DESCRIPTION:
It is estimated that between 1.5% and 7.5% of children experience encopresis. In most children, encopresis is a complication of long-standing constipation. Encopresis is defined as the repeated passage of feces in inappropriate places at least once a month, for three months, and not induced through substances or due to a general medical condition. Typically, treatment consists of medical management alone, which focuses on diet and/or laxative therapy and has a relatively low success rate. A combination of specialized medical and behavioral interventions for encopresis (Enhanced Toilet Training) has been found to have high success rates. Unfortunately, it is not readily available because of a lack of trained professionals to deliver the treatment and the amount of time and costs spent in delivering this treatment. Internet interventions, however, may lower some of the barriers associated with traditional face-to-face treatments by removing the inconvenience of scheduling appointments, missing work/school, and traveling to and from a clinician's office. This study will evaluate whether an Internet intervention is more effective than patient education in treating pediatric encopresis. This study will also evaluate whether stepped care support is additive to the effectiveness of the Internet intervention. Stepped care will involve adding personal e-mail and phone support to help families overcome obstacles to using and implementing the intervention.

Participants are randomized to receive a patient education website, the Internet intervention alone, or the Internet intervention plus stepped care. The intervention period lasts for 6 weeks. During the intervention period, subjects assigned to the patient education website will be given content addressing treatment of encopresis. Those assigned to use the Internet intervention will review interactive tutorials tailored to the user's difficulties. The stepped care group will receive the Internet intervention as well as additional support if they fail to reach specific intervention milestones. All families will complete assessment questionnaires and daily diaries of the children's symptoms and bowel behaviors for one week at baseline, following the intervention period, and at 6 and 12 months follow-up.

ELIGIBILITY:
Criteria for inclusion:

A child and his or her parent/caregiver may participate in the study if:

* The parent/caregiver is the legal guardian of his or her child.
* The child is between the ages of 5 and 12.
* The child has had fecal accidents for at least the past three months.
* The child has had at least two fecal accidents during the past two weeks.
* The child and parent/caregiver have regular access to the Internet, either through the family computer or another readily accessible computer.

Criteria for exclusion:

A child and his or her parent/caregiver may not participate in the study if:

* The child has had an Endorectal Pull-Through Procedure.
* The child has a history of Short Bowel Syndrome.
* The child has a diagnosis of a primary illness responsible for fecal soiling (e.g., Spinal Bifida, Hirschsprung's Disease).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Primary encopretic symptoms (as defined by): 1. Number of episodes of fecal soiling 2. Number of bowel movements in the toilet 3. Increased trips to the bathroom (both parent and self-prompted) | Baseline, 6 weeks, 6 months, 1 year

SECONDARY OUTCOMES:
Behavior change around encopresis (as measured by): 1. Appropriate clean-out 2. Appropriate laxative use 3. Appropriate rectus abdominis straining 4. Toileting routine | Baseline, 6 weeks, 6 months, 1 year
Secondary encopretic symptoms (as defined by): 1. Appropriate bowel movement consistency 2. Reduced bowel-specific difficulties | Baseline, 6 weeks, 6 months, 1 year
Frequency and Severity of perianal pain | Baseline, 6 weeks, 6 months, 1 year
Costs (as measured by): 1. Time spent managing symptoms 2. Doctor visits 3. Medication usage 4. Missed school/work days 5. Diapers used 6. Therapist time in stepped-care component 7. Expenses associated with building and maintaining web program | Baseline, 6 weeks, 6 months, 1 year
Website Utilization (as measured by): 1. Time spent on website 2. Number of log-ins 3. Number of completed website Modules and Follow-Ups | Throughout Intervention (from Baseline to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Ritterband, PhD, Principal Investigator — University of Virginia Health Systems
Locations (1):
- University of Virginia Health System, Department of Psychiatry and Neurobehavioral Sciences, Behavioral Health and Technology, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Ritterband LM, Cox DJ, Walker LS, Kovatchev B, McKnight L, Patel K, Borowitz S, Sutphen J. An Internet intervention as adjunctive therapy for pediatric encopresis. J Consult Clin Psychol. 2003 Oct;71(5):910-7. doi: 10.1037/0022-006X.71.5.910. PMID 14516239
- [Background] Cox DJ, Morris JB Jr, Borowitz SM, Sutphen JL. Psychological differences between children with and without chronic encopresis. J Pediatr Psychol. 2002 Oct-Nov;27(7):585-91. doi: 10.1093/jpepsy/27.7.585. PMID 12228330
- [Background] Ritterband LM, Thorndike F. Internet interventions or patient education web sites? J Med Internet Res. 2006 Sep 29;8(3):e18; author reply e19. doi: 10.2196/jmir.8.3.e18. No abstract available. PMID 17032634
- [Background] Ritterband LM, Borowitz S, Cox DJ, Kovatchev B, Walker LS, Lucas V, Sutphen J. Using the internet to provide information prescriptions. Pediatrics. 2005 Nov;116(5):e643-7. doi: 10.1542/peds.2005-0404. PMID 16263978
- [Background] Borowitz SM, Cox DJ, Kovatchev B, Ritterband LM, Sheen J, Sutphen J. Treatment of childhood constipation by primary care physicians: efficacy and predictors of outcome. Pediatrics. 2005 Apr;115(4):873-7. doi: 10.1542/peds.2004-0537. PMID 15805358
- [Background] Cox DJ, Ritterband LM, Quillian W, Kovatchev B, Morris J, Sutphen J, Borowitz S. Assessment of behavioral mechanisms maintaining encopresis: Virginia Encopresis-Constipation Apperception Test. J Pediatr Psychol. 2003 Sep;28(6):375-82. doi: 10.1093/jpepsy/jsg027. PMID 12904449
- [Background] Borowitz SM, Cox DJ, Tam A, Ritterband LM, Sutphen JL, Penberthy JK. Precipitants of constipation during early childhood. J Am Board Fam Pract. 2003 May-Jun;16(3):213-8. doi: 10.3122/jabfm.16.3.213. PMID 12755248